CLINICAL TRIAL: NCT05507801
Title: The Effect of Protein on Appetite and Food Intake in More and Less Active Older Adults.
Brief Title: Protein and Satiety in Older Adults (PROSAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Ministry of National Education, Turkey (Other Government)
Responsible Party: Principal Investigator, Miriam Clegg, Associate Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UREC 21/40
Record Dates: First submitted 2022-08-11; First posted 2022-08-19 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Appetitive Behavior; Gastric Emptying; Physical Activity; Energy Intake
Keywords: protein; physical activity; older adults; appetite; energy intake; satiety
MeSH Terms: conditions — Appetitive Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Physically Active Group (Experimental): Based on accelerometer data, women with 162 ≥ min/per day moderate and vigorous activity or men 133.25 ≥ min/per day moderate and vigorous activity.
  Interventions: Other: High Protein Milkshake; Other: Normal Milkshake
- Low Physically Active Group (Experimental): Based on accelerometer data, women with 108.25 ≤ min/per day moderate and vigorous activity or men 100.1 ≤ min/per day moderate and vigorous activity.
  Interventions: Other: High Protein Milkshake; Other: Normal Milkshake

INTERVENTIONS:
Other: High Protein Milkshake — A milkshake with high protein level; including whey protein, fat free strawberry yogurt and whole milk - 337 kcal, 27 g carbohydrate, 57 g protein, 16 g fat.
Other: Normal Milkshake — A milkshake with normal protein level; including nesquik (strawberry), fat free strawberry yogurt, whole milk, double cream, whey protein and sweetener - 331 kcal, 64 g carbohydrate, 17 g protein, 19 g fat.

SUMMARY:
This study aims to assess the effect of protein on appetite, food intake and gastric emptying in older adults (≥ 65 years) that are more and less active.

DETAILED DESCRIPTION:
To investigate the differences in food intake in older adults that are more or less active and assess any differential responses to protein intake.

To compare the effect of meals with high or low protein level but equal in energy and volume on appetite and gastric emptying in older adults that are more or less active (≥ 65 years).

ELIGIBILITY:
Inclusion Criteria:

* healthy
* aged ≥ 65 years

Exclusion Criteria:

* having diabetes or disability or any disease that are likely to influence physical activity or appetite.
* having an allergy to any of the test foods;
* disliking or cannot eat any of the test foods;
* being obese (BMI > 30 kg/m2);
* taking medications known to influence appetite, food intake or body weight in the past three months;
* being on a weight loss diet;
* smoking more than 10 cigarettes a day;
* not meeting the cut-off point criteria based on the accelerometer data (108.25 ≤ min/per day of moderate and vigorous activity for women or 162 ≥ min/per day moderate and vigorous activity for women and 100.1 ≤ min/per day of moderate and vigorous activity for men or 133.25 ≥ min/per day moderate and vigorous activity for men).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Ad-libitum meal consumption | 2 days in total
  Consumption of the ad-libitum meal is measured (g). Participants are instructed to eat until they feel comfortable full and are given 20 min to consume the meal.

SECONDARY OUTCOMES:
Ratings of appetite | 2 days in total
  Appetite are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100).
Gastric Emptying | 2 days in total
  Gastric emptying is measured using of 100 microliters of 13C Octanoic Acid breath test
Ratings of palatability | 2 days in total
  Palatability ratings are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however, it is possible that some of the individual (unliked / non-identifiable) data will be useful in a meta-analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] Morell P, Fiszman S. Revisiting the role of protein-induced satiation and satiety. Food Hydrocolloids. 2017 Jul 1;68:199-210.
- [Background] Timiras PS. Physiological basis of aging and geriatrics, CRC Press. 2022
- [Background] Ahmed T, Haboubi N. Assessment and management of nutrition in older people and its importance to health. Clin Interv Aging. 2010 Aug 9;5:207-16. doi: 10.2147/cia.s9664. PMID 20711440
- [Background] St-Onge MP, Gallagher D. Body composition changes with aging: the cause or the result of alterations in metabolic rate and macronutrient oxidation? Nutrition. 2010 Feb;26(2):152-5. doi: 10.1016/j.nut.2009.07.004. Epub 2009 Dec 8. PMID 20004080
- [Background] Margetts BM, Thompson RL, Elia M, Jackson AA. Prevalence of risk of undernutrition is associated with poor health status in older people in the UK. Eur J Clin Nutr. 2003 Jan;57(1):69-74. doi: 10.1038/sj.ejcn.1601499. PMID 12548299
- [Background] Giezenaar C, Trahair LG, Luscombe-Marsh ND, Hausken T, Standfield S, Jones KL, Lange K, Horowitz M, Chapman I, Soenen S. Effects of randomized whey-protein loads on energy intake, appetite, gastric emptying, and plasma gut-hormone concentrations in older men and women. Am J Clin Nutr. 2017 Sep;106(3):865-877. doi: 10.3945/ajcn.117.154377. Epub 2017 Jul 26. PMID 28747330
- See also: Healthy eating overview-Maintaining a healthy weight. — https://www.ageuk.org.uk/globalassets/age-ni/documents/information-guides/ageukig38_healthy_eating_inf.pdf
- See also: Exercise as you get older. — http://www.nhs.uk/live-well/exercise/